CLINICAL TRIAL: NCT02909855
Title: Factors Associated With Parental Observation of Side Effects Following the Child Flu Vaccine
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/LO/1003
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Influenza Vaccine, Influenza
Keywords: children; psychological predictors; side-effects; vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Parents of children aged 2-4 who will receive the child flu vaccine from their general practitioner (GP)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Participants in this study will not receive any interventions as part of the study.

SUMMARY:
This study investigates whether there are psychological predictors of parental perception of side-effects following vaccination with the child flu vaccine. We will also investigate whether the perception of side-effects affects parents' intention to vaccinate their child again in the following flu season, as well as whether there are underlying differences in parents' cognitive biases between those who do and do not re-vaccinate their child.

DETAILED DESCRIPTION:
In 2012, the British Joint Committee on Vaccination and Immunisation (JCVI) recommended that the influenza vaccination programme be extended to include children aged 2 to 16. In the three flu seasons in which the child flu immunisation programme has been running (2013-14, 2014-15, 2015-16), uptake rates have been low (approximately 40%). Multiple factors are likely to underlie the poor uptake, including thinking the vaccine was unsafe and ineffective and having experienced side-effects related to the vaccine previously.

Although symptoms are commonly reported following vaccinations, their causes are not always straightforward. Although a minority may be directly attributable to the vaccine itself, others may reflect pre-existing or coincidental symptoms that are misattributed to the vaccine. Following vaccination, an expectation that the vaccine causes side-effects may also contribute to parents detecting symptoms in their child that might otherwise have gone unnoticed. Perception of side-effects may also influence the parent's decision to vaccinate their child again in following years.

Other possible factors influencing parents' perception of side-effects and their willingness to vaccinate their child again are their personal health beliefs and their interpretations of the information they are given about vaccination and side-effects. These cognitive processes can be measured objectively using experimental tasks, and can reveal characteristic patterns, or 'cognitive biases' which govern behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Parents of guardians of children aged 2-4 on 31st August 2016 (i.e. born September 1st 2011 to August 31st 2014) who receive the flu vaccine at the GP
* Parents must be aged 18 or over
* Parents must be fluent in English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Parents of guardians of children aged 2-4 on 31st August 2016 (i.e. born September 1st 2011 to August 31st 2014) who receive the flu vaccine at the GP
  * Parents must be aged 18 or over
  * Parents must be fluent in English
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of participants who perceive their child to have treatment-related adverse events from the child flu vaccine | October 2016 - March 2017
  Using questionnaire materials as a method of assessment

SECONDARY OUTCOMES:
Intention to re-vaccinate child | October 2016 - March 2017
  Using a scale as a method of assessment
Negative interpretative bias scores as assessed by the scrambled sentences and similarity ratings tasks | October 2016 - March 2017

OTHER OUTCOMES:
Vaccination status of child for flu at end of 2017/18 flu season | January - March 2018

CONTACTS AND LOCATIONS:
Overall Officials: G James Rubin, PhD, Principal Investigator — King's College London
Locations (11):
- United Kingdom (11):
  - Albion Street Group Practice, London
  - Claremont Medical Centre, London
  - Herne Hill Group Practice, London
  - Honor Oak Group Practice, London
  - Hurley Clinic, London
  - Links Medical Practice, London
  - Morden Hall Medical Centre, London
  - Park Group Practice, London
  - Paxton Green Group Practice, London
  - The Rosendale Surgery, London
  - Woodlands Practice, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith LE, Amlot R, Weinman J, Yiend J, Rubin GJ. Why do parents not re-vaccinate their child for influenza? A prospective cohort study. Vaccine. 2020 Jun 2;38(27):4230-4235. doi: 10.1016/j.vaccine.2020.04.029. Epub 2020 May 5. PMID 32386745
- [Derived] Smith LE, Weinman J, Amlot R, Yiend J, Rubin GJ. Parental Expectation of Side Effects Following Vaccination Is Self-fulfilling: A Prospective Cohort Study. Ann Behav Med. 2019 Mar 1;53(3):267-282. doi: 10.1093/abm/kay040. PMID 29868792